CLINICAL TRIAL: NCT06279988
Title: BRING-UP 3 Heart Failure
Acronym: BRING-UP3HF
Status: Recruiting | Type: Observational
Sponsor: Heart Care Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: K24
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational study is to assess the level of adherence to guideline recommendations regarding the management of patients with Heart Failure with Reduced Ejection Fraction (HFrEF); - the safety profile of the implementation of recommended treatments; - to monitor treatment patterns of patients with acute hert failure (HF); - to monitor treatment patterns of all patients with chronic HF irrespective of the level of ejection fraction (EF).

DETAILED DESCRIPTION:
Observational, prospective, multicenter study conducted in a large, representative sample of Italian cardiology centers.

Phases 1:

1. First educational intervention to discuss the recommendations of guidelines and treatment patterns in specific phenotypes of patients.
2. Data collection for 3 months or up to 30 consecutive patients with chronic HF or acute HF (both de novo and worsening).
3. Evaluation of the primary and secondary end-points of the study at 6 months after enrollment. Modifications of treatments will be monitored during the 6 months follow-up.
4. Second educational intervention to share the results of the first enrollment period of the study focusing the attention on existing gaps between guidelines recommendations and clinical practice.
5. New data collection for other 3 months or up to 30 consecutive patients with chronic HF or acute HF (both de novo and worsening).
6. Additional evaluation of the primary and secondary end-points of the study at 6 months after enrollment. Modifications of treatments will be monitored during the 6 months follow-up.
7. 12-month follow-up for all patients included in both enrolment phases of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. Males and females at birth.
3. Any ejection fraction level (level of ejection fraction measured in the 6 months preceding enrollment).
4. Ambulatory chronic HF or Hospitalized de-novo or worsening HF.
5. Signed informed consent

Diagnosis will be made by the local attending physician following the ESC guidelines recommendations.

Exclusion Criteria:

1. Active neoplasia or very severe disease compromising short-medium term life expectancy.
2. Participation in interventional studies.
3. Patients already enrolled into the study from another participating center or in the previous enrolling phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with chronic HF and those admitted for acute (de novo or worsening) HF.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Rate of adherence to Guideline-Directed Medical Therapy (GDMTs) in HFrEF | 6 months
  To assess the rate of patients with HFrEF appropriately treated with the 4 therapeutic pillars [Angiotensin Converting Enzyme Inhibitors (ACE-i)/Angiotensin Receptor Blockers (ARBs)/Angiotensin Receptor/Neprilysin Inhibitor (ARNI), betablockers, mineralocorticoid receptor antagonist (MRAs), Sodium-Glucose Co-Transporter-2 (SGLT2i)] recommended by current European Society of Cardiology (ESC) 2021 guidelines. Patients with a documented contraindication to one or more of the 4 recommended therapeutic pillars will be included in the group of appropriately treated patients.

SECONDARY OUTCOMES:
Rate of patient achieving appropriate dosages of GDMTs | 6 months
  to assess the rate of patients treated with appropriate dosages* of:ACE-i/ARBs/ARNI, betablockers, MRAs, SGLT2i and to describe and assess the rate of adverse reactions reported by the Investigators when detected during their usual clinical practice
  *For the purpose of the present study appropriate dosage is defined as a dosage ≥50% of the maximal recommended dosage by the current guidelines
Treatment patterns of patients with Heart failure with mildly reduced ejection fraction (HFmrEF) and Heart failure with preserved ejection fraction (HFpEF) | 6 months
  To assess how novel treatment recommendations for HFmrEF and HFpEF are implemented in practice, specifically the rate of use of ARNI and SGLT2i and to describe and assess the rate of adverse reactions reported by the Investigators when detected during their usual clinical practice
Treatment patterns of patients with Acute Heart Failure (AHF) irrespective of the level of EF | 6 months
  To assess the rate of use of vasopressors, vasodilators, renal replacement therapy and mechanical circulatory support, pharmacological treatments and follow-up planning at discharge and to describe and assess the rate of adverse reactions reported by the Investigators when detected during their usual clinical practice.
All cause and specific causes of death and hospitalization (Exploratory endpoint) | 12 months
  To evaluate the rate of occurrence of clinical events during the 12 months follow-up of each enrolment phase. Specifically all-cause death, all-cause hospitalizations, specific causes of death and hospitalizations.

CONTACTS AND LOCATIONS:
Locations (187):
- Italy (187):
  - Ospedale Santo Spirito - Sc Cardiologia, Casale Monferrato, AL
  - Ospedale San Giacomo - Sc Cardiologia, Novi Ligure, AL
  - Ospedali Riuniti - Sod Cardiologia Ospedaliera E Utic, Ancona, AN
  - Irccs Inrca - Uo Cardiologia/Utic/Telecardiologia, Ancona, AN
  - Ospedale San Donato - U.O.C Cardiologia, Arezzo, AR
  - Ospedale Valdichiana Santa Margherita - Uosd Cardiologia S.O. Cortona, Cortona, AR
  - Aorn San Giuseppe Moscati - U.O. Cardiologia/Utic 'D. Rotiroti', Avellino, AV
  - Ospedale Miulli - U.O.C. Cardiologia - Utic, Acquaviva delle Fonti, BA
  - Ospedale Della Murgia - Fabio Perinei - S.C. Cardiologia-Utic, Altamura, BA
  - Ospedale San Paolo - Cardiologia-Utic, Bari, BA
  - Ics Maugeri Spa Societa' Benefit Irccs Bari - Cardiologia Riabilitativa, Bari, BA
  - Mater Dei Hospital - Riabilitazione Cardiologica, Bari, BA
  - Ospedale Di Venere - U.O.C. Di Cardiologia, Carbonara di Bari, BA
  - Ospedale San Giacomo - Uoc Cardiologia, Monopoli, BA
  - Ospedale Degli Infermi - Sc Di Cardiologia, Ponderano, BI
  - Presidio Ospedaliero "Santa Maria Del Prato" - U.O.C. Di Cardiologia-Utic, Feltre, BL
  - Ospedale Di Bentivoglio - U.O. Cardiologia Pianura, Bentivoglio, BO
  - Ospedale Maggiore - U.O.C. Di Cardiologia, Bologna, BO
  - Ospedale Policlinico S. Orsola-Malpighi - Medicina Interna - Borghi, Bologna, BO
  - Ospedale Perrino - U.O.C. Di Cardiologia, Brindisi, BR
  - Istituto Ospedaliero Fondazione Poliambulanza - Unita Operativa Di Cardiologia E Utic, Brescia, BS
  - Ospedale Di Desenzano Del Garda - Divisione Di Cardiologia - U.C.C., Desenzano del Garda, BS
  - Ospedale Civile 'La Memoria' - U.O. Di Cardiologia, Gavardo, BS
  - Istituti Clinici Scientifici Maugeri Irccs Sede Di Lumezzane - U.O. Di Cardiologia Riabilitativa, Lumezzane, BS
  - Ospedale Monsignor Angelo R. Di Miccoli - Uoc Cardiologia/Utic, Barletta, BT
  - Ospedale Caduti in Guerra - U.O.S.V.D Di Riabilitazione Cardiologica, Canosa di Puglia, BT
  - Ospedale Centrale Bolzano - Cardiologia E Prove Funzionali, Bolzano, BZ
  - Azienda Ospedaliera S. Anna E S. Sebastiano - U.O. Cardiologia D'Emergenza Con Utic, Caserta, CE
  - Villa Delle Magnolie - Riabilitazione Cardiologica, Castel Morrone, CE
  - Casa Di Cura San Michele - Uo Cardiologia, Maddaloni, CE
  - Ospedale Policlinico Ss. Annunziata - Uoc Cardiologia-Utic, Chieti, CH
  - Azienda Ospedaliera Santa Croce E Carle - Sc Cardiologia, Cuneo, CN
  - Ospedale Regina Montis Regalis - U.O. Cardiologia-Utic, Mondovì, CN
  - Ospedale Maggiore Ss. Annunziata - Sc Cardiologia, Savigliano, CN
  - Ospedale Pietro E Michele Ferrero - Cardiologia E Utic, Verduno, CN
  - Ospedale S. Anna - U.O.C. Di Cardiologia, San Fermo della Battaglia, CO
  - Ospedale Oglio Po - U.O. Di Cardiologia-Utic, Casalmaggiore, CR
  - Ospedale Civile Ferrari - U.O.C. Cardiologia-Utic, Castrovillari, CS
  - Ospedale Spoke Paola- Cetraro Po Paola - Utic Cardiologia, Paola, CS
  - P.O. Garibaldi-Nesima - Arnas Garibaldi - U.O.C. Di Cardiologia Con Utic, Catania, CT
  - Policlinico Catania Po G. Rodolico - Cardiologia Utic, Catania, CT
  - Azienda Ospedaliera Cannizzaro - Uoc Cardiologia, Catania, CT
  - P.O. "Materdomini" - A.O.U. "Renato Dulbecco" - Ssd Cardiologia Riabilitativa, Catanzaro, CZ
  - P.O. "Pugliese" - A.O.U. "Renato Dulbecco" - Utic-Emodinamica E Cardiologia Interventistica, Catanzaro, CZ
  - Presidio Ospedaliero Umberto I - Cardiologia - Utic- Riabilitazione, Enna, EN
  - Ospedale G.B. Morgagni - L. Pierantoni - U.O. Cardiologia, Forlì, FC
  - Ospedale Ss. Annunziata - U.O. Di Cardiologia Provinciale, Cento, FE
  - Arcispedale Sant'Anna - U.O. Cardiologia, Ferrara, FE
  - Ospedale Del Delta - U.O. Cardiologia, Lagosanto, FE
  - Policlinico Riuniti - S.C. Di Cardiologia Universitaria-Utic, Foggia, FG
  - Ospedale Casa Sollievo Della Sofferenza - Cardiologia - Utic - Riabil Cardiologica, San Giovanni Rotondo, FG
  - Ospedale San Giuseppe - Cardiologia, Empoli, FI
  - Ospedale Santa Maria Nuova - Cardiologia, Florence, FI
  - Ospedale San Giovanni Di Dio - Sos Cardiologia, Florence, FI
  - Aou Careggi - Geriatria - Utig, Florence, FI
  - Ospedale Padre Antero Micone - Sc Cardiologia - Utic, Genova, GE
  - Irccs Ospedale Policlinico San Martino - Clinica Malattie Apparato Cardiovascolare, Genova, GE
  - Ospedale Del Tigullio Polo Lavagna - Sc Cardiologia E Utic, Lavagna, GE
  - Ospedale San Giovanni Di Dio - Sc Cardiologia (Gorizia-Monfalcone), Gorizia, GO
  - Ospedale Civile San Polo - Sc Cardiologia (Gorizia-Monfalcone), Monfalcone, GO
  - Ospedale S. Andrea - Alta Maremma - Uosd Cardiologia, Massa Marittima, GR
  - Ospedale Alessandro Manzoni - S.C. Di Cardiologia, Lecco, LC
  - Ospedale San Giuseppe Da Copertino - U.O. Di Cardiologia, Copertino, LE
  - Ospedale Vito Fazzi - Uoc Cardiologia-Utic Ed Emodinamica, Lecce, LE
  - Ospedale Ignazio Veris Delli Ponti - Uoc Cardiologia-Utic "E. Vilei", Scorrano, LE
  - Ospedali Riuniti - U.O.C. Cardiologia E Utic, Livorno, LI
  - Ospedale Villamarina - Cardiologia E Utic Piombino Elba, Piombino, LI
  - Nuovo Ospedale Versilia - Sc Cardiologia, Camaiore, LU
  - Ospedale Santa Croce - Uosd Cardiologia E Di Continuita Assist., Castelnuovo di Garfagnana, LU
  - Ospedale Pio Xi - U.O.C. Di Cardiologia, Desio, MB
  - Policlinico Di Monza - Cardiologia Clinica E Utic, Monza, MB
  - Nuovo Ospedale Di Vimercate - S.C. Cardiologia E Utic, Vimercate, MB
  - Ospedale Generale Provinciale - U.O. Cardiologia, Macerata, MC
  - Irccs Centro Neurolesi Bonino Pulejo - P.O Piemonte - Cardiologia E Utic, Messina, ME
  - Azienda Ospedaliera Papardo - U.O. Cardiologia Con Utic - Emodinamica, Messina, ME
  - Asst Papa Giovanni Xxiii - Sc Cardiologia 1, Bergamo, MI
  - Ospedale Di Cernusco Sul Naviglio - U. O. Di Cardiologia E Ucc, Cernusco sul Naviglio, MI
  - Ospedale Edoardo Bassini - Sc Cardiologia-Ucc Asst Nord Milano (Bassini-Ssg), Cinisello Balsamo, MI
  - Asst Ovest Milanese - Po Di Legnano - Cardiologia E Unita' Coronarica, Legnano, MI
  - Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico - Uoc Malattie Cardiovascolari, Milan, MI
  - Ospedale Fatebenefratelli E Oftalmico - Cardiologia E U.C.C., Milan, MI
  - Centro Cardiologico Monzino Irccs - Scompenso,Cardiologia Clinica, Milan, MI
  - Istituti Clinici Scientifici Maugeri Irccs Sede Di Milano - Riabilitazione Cardiologica, Milan, MI
  - Istituti Clinici Scientifici Maugeri Irccs Sede Di Milano - Uo Cure Subacute, Milan, MI
  - ASST SANTI PAOLO E CARLO - PO San Carlo - CARDIOLOGIA-UCC, Milan, MI
  - Irccs Ospedale Galeazzi - Sant'Ambrogio - Cardiologia Universitaria Ed Imaging Cardiaco, Milan, MI
  - Asst Ospedale Metropolitano Niguarda - Cardiologia 2 - Insufficienza Cardiaca E Trapianto, Milan, MI
  - Clinica San Carlo - U.O. Cardiologia-Unita'Cure Coronariche, Paderno Dugnano, MI
  - Presidio Ospedaliero Di Passirana - Cardiologia Riabilitativa, Passirana, MI
  - Istituto Clinico Humanitas - Irccs - Cardiologia Clinica, Interventistica E Ucc, Rozzano, MI
  - Irccs Policlinico San Donato - U.O. Cardiologia Con Utic, San Donato Milanese, MI
  - Irccs Policlinico Multimedica - Uo Di Cardiologia, Sesto San Giovanni, MI
  - Ospedale Madonna Delle Grazie - Ssd Utic, Matera, Mount
  - Ospedale Giovanni Paolo Ii - Uosd Utic, Policoro, Mount
  - Ospedale Santa Maria Bianca - U.O. Di Cardiologia, Mirandola, MO
  - Ospedale Di Sassuolo - Cardiologia, Sassuolo, MO
  - Ospedale Giovanni Paolo Ii - Utic - Cardiologia, Olbia, OT
  - Fondazione G. Giglio - U.O. Di Cardiologia, Cefalù, PA
  - Ospedale Buccheri La Ferla Fatebenefratelli - Ssd Riabilitazione Cardiovascolare, Palermo, PA
  - Arnas P.O. Civico E Benfratelli - Uoc Utic, Palermo, PA
  - Arnas P.O. Civico E Benfratelli - Uosd Cardiologia Clinica Trattam. Scompenso Card., Palermo, PA
  - Maria Eleonora Hospital - Cardiologia, Palermo, PA
  - Aor Villa Sofia-Cervello P.O. Cervello - U.O. Cardiologia - Cervello, Palermo, PA
  - Aor Villa Sofia-Cervello Po Villa Sofia - Uoc Cardiologia E Utic E Emodinamica -Villa Sofia, Palermo, PA
  - Ospedale Unico Della Val Tidone - Cardiologia E Riabilitazione, Castel San Giovanni, PC
  - Ospedale Civile 'Guglielmo Da Saliceto' - Uoc Cardiologia E Utic, Piacenza, PC
  - Ospedali Riuniti Padova Sud - U.O.C. Cardiologia, Monselice, PD
  - Ospedale Civile Dello Spirito Santo - Cardiologia Con Utic, Pescara, PE
  - Presidio Ospedaliero Citta' Di Castello - U.O. Cardiologia/Utic, Città di Castello, PG
  - Nuovo Ospedale San Giovanni Battista - S.C. Cardiologia, Foligno, PG
  - Ospedale Gubbio-Gualdo Tadino - U.O. Di Utic E Cardiologia, Gubbio, PG
  - Centro Servizi Grocco - Cardiologia Riabilitativa E Prevenzione, Perugia, PG
  - Ftgm - Stabilimento Di Pisa - Cardiologia E Medicina Cardiovascolare, Pisa, PI
  - Ospedale Generale Provinciale Lotti - U.O. Malattie Cardiovascolari Vde E Avc, Pontedera, PI
  - Ospedale Di S. Vito Al Tagliamento - Ssd Cardiologia San Vito - Spilimbergo, San Vito al Tagliamento, PN
  - Ospedale San Jacopo - Soc Cardiologia, Pistoia, Point
  - Ospedale Civile - U.O.C. Cardiologia - Utic, Fidenza, PR
  - Fondazione Irccs Policlinico San Matteo - Uoc Cardiologia 1, Pavia, PV
  - Istituti Clinici Scientifici Maugeri Irccs Sede Di Pavia - U.O. Di Riabilitazione Cardiologica, Pavia, PV
  - Ospedale Civile - U.O. Di Cardiologia, Voghera, PV
  - Ospedale Civile - Uo Servizio Cardiologia, Lugo, RA
  - Ospedale Civile Santa Maria Delle Croci - Uoc Cardiologia, Ravenna, RA
  - Ospedale Civile Di Guastalla - Sos Cardiologia E Riabilitazione Card Area Nord, Guastalla, RE
  - Po Santa Maria Nuova - Ausl Re Irccs - Soc Cardiologia Ospedaliera, Reggio Emilia, RE
  - Ospedale Riccardo Guzzardi - U.O.C. Di Cardiologia-Utic, Vittoria, RG
  - P.O. San Camillo de Lellis - U.O.C. Cardiologia, Rieti, RI
  - Ospedale Dei Castelli - U.O.C. Di Cardiologia E Utic, Ariccia, RM
  - Ospedale Civile San Paolo - U.O.C. Cardiologia - Utic, Civitavecchia, RM
  - Campus Biomedico - Cardiologia, Roma, RM
  - P.O. San Filippo Neri - Asl Roma 1 - Cardiologia Clinica E Riabilitativa, Roma, RM
  - Inmi Lazzaro Spallanzani Irccs - Servizio Di Cardiologia Del Dipartimento Clinico, Roma, RM
  - Ospedale San Camillo - Uoc Cardiologia, Roma, RM
  - Ospedale Sandro Pertini - Uoc Cardiologia, Roma, RM
  - Policlinico Casilino - U.O.C. Cardiologia, Roma, RM
  - Ao San Giovanni Addolorata - Uoc Cardiologia D'Urgenza E Utic, Roma, RM
  - Ospedale Isola Tiberina - Uoc Cardiologia Diagnostica Interventistica-Utic, Roma, RM
  - Ospedale Sant'Andrea Di Roma - U.O.C. Cardiologia, Roma, RM
  - Ospedale Santo Spirito - Uoc Cardiologia, Roma, RM
  - Ospedale San Giovanni Evangelista - U.O.C. Di Cardiologia - Utic, Tivoli, RM
  - Ospedale Infermi - U.O. Cardiologia, Rimini, RN
  - Ospedale Maria Ss. Addolorata - U.O. Di Cardiologia Utic, Eboli, SA
  - Aou S. Giovanni Di Dio-Ruggi D'Aragona - Cardiologia Intensiva Ospedaliera, Salerno, SA
  - Aou S. Giovanni Di Dio-Ruggi D'Aragona - Ssd Utic, Salerno, SA
  - Ospedale San Luca - U.O. Utic - Cardiologia, Vallo della Lucania, SA
  - Ospedale Dell'Alta Val D'Elsa - Uosd Cardiologia-Utic, Poggibonsi, SI
  - Aou Senese Ospedale S. Maria Alle Scotte - Cardiologia, Siena, SI
  - Ospedale San Bartolomeo - Sc Riabilitazione Cardiologica, Sarzana, SP
  - Ospedale E. Muscatello - U.O. Di Cardiologia - Utic, Augusta, SR
  - Ospedale G. Di Maria - Cardiologia Utic, Avola, SR
  - Ospedale Ss. Annunziata - Cardiologia Clinica Ed Interventistica, Sassari, SS
  - Ospedale Nostra Signora Di Bonaria - U.O.C. Cardiologia E Utic, San Gavino Monreale, SU
  - Po Ponente - Ospedale Santa Corona - Sc Cardiologia Ponente, Pietra Ligure, SV
  - P.O. Levante - Ospedale San Paolo - S.C. Cardiologia Levante, Savona, SV
  - Casa Di Cura Villa Verde - Cardiologia, Taranto, TA
  - Ospedale Santa Chiara - Divisione Di Cardiologia, Trento, TN
  - Ospedale Civico - Sc Cardiologia, Chivasso, TO
  - Por Cirié- Lanzo Presidio Cirié - S.C. Cardiologia, Cirié, TO
  - Ospedale Civile - S.C. Cardiologia, Ivrea, TO
  - Aou San Luigi Gonzaga - S.C.D.O. Cardiologia, Orbassano, TO
  - Aou Citta' Della Salute E Della Scienza - S.C. Cardiologia U, Torino, TO
  - Ospedale Martini - Cardiologia (Mrt-Mv), Torino, TO
  - Ospedale Maria Vittoria - Cardiologia (Mrt-Mv), Torino, To
  - Ospedale San Giovanni Bosco - Sc Cardiologia, Torino, TO
  - Ospedale Santa Maria Del Carmine - Cardiologia, Rovereto, Trento
  - Asugi Trieste - Sc Patologie Cardiovascolari, Trieste, TS
  - Pou "Santa Maria Della Misericordia" - S.O.C. Cardiologia, Udine, UD
  - Ospedale Multimedica Castellanza - Cardiologia, Castellanza, VA
  - Presidio Ospedaliero Di Saronno - U.O.C. Di Cardiologia, Saronno, VA
  - Ospedale Di Circolo Galmarini - Cardiologia, Tradate, VA
  - Ospedale Sant'Andrea - Sc Cardiologia, Vercelli, VC
  - Ospedale Dell'Angelo - U.O.C. Cardiologia, Mestre, VE
  - Ospedale P.F. Calvi - Uos Di Cardiologia Riabilitativa, Noale, VE
  - Ospedale Civile - U.O.C. Di Cardiologia, Arzignano, VI
  - Ospedale Alto Vicentino - U.O.C. Cardiologia - Ucic, Santorso, VI
  - Ospedale G. Fracastoro - U.O.C. Di Cardiologia, San Bonifacio, VR
  - Ospedale Civita Castellana - Ssd Cardiologia, Civita Castellana, VT
  - Ospedale Belcolle - Uoc Cardiologia Ed Emodinamica, Viterbo, VT
  - Ospedale Ss. Trinita' - S.C. Di Cardiologia, Borgomanero
  - Istituti Clinici Scientifici Maugeri Irccs Sede Di Veruno - Uo Cardiologia Riabilitativa, Gattico
  - Ospedale Anna Rizzoli - Cardiologia-Utic, Lacco Ameno
  - Ospedale Buon Consiglio Fatebenefratelli - U.O.Complessa Di Cardiologia E Utic, Napoli
  - Aorn Cardarelli - U.O. Cardiologia Con Utic, Napoli
  - Aorn Ospedale Dei Colli - P.O. Monaldi - Uosd Card. Riabilitativa Intensiva E Scompenso, Napoli
  - Aorn Ospedale Dei Colli - P.O. Monaldi - Uosd Malattie Cardiologiche Congenite Adulti-Guch, Napoli
  - Ospedale S. Giovanni Bosco - Sc Cardiologia - Utic, Napoli
  - Aou Maggiore Della Carita' - Scdo Cardiologia Ii, Novara
  - Ospedale Santa Maria Delle Grazie - U.O. Cardiologia - Utic Con Emodinamica, Pozzuoli

REFERENCES:
- [Derived] Basile C, Oliva F, Orso F, Colivicchi F, Cipriani MG, Di Lenarda A, Gori M, Gorini M, Iacoviello M, Marini M, Gabrielli D, Maggioni AP. Age- and Sex-related Differences in Heart Failure Characteristics and Treatment Patterns Across the Ejection Fraction Spectrum: First Data from the BRING-UP-3 Heart Failure Study. Eur Heart J Qual Care Clin Outcomes. 2025 Sep 24:qcaf113. doi: 10.1093/ehjqcco/qcaf113. Online ahead of print. PMID 40987455
- [Derived] Oliva F, Orso F, Colivicchi F, Cipriani MG, DI Lenarda A, Gabrielli D, Gori M, Gorini M, Iacoviello M, Lucci D, Marini M, Amico F, Bertoli D, Carigi S, D'Elia E, DI Fusco SA, Fucili A, Lanati G, Menegato A, Moretti M, Navazio A, Passantino A, Pulignano G, Ruzzolini M, Scardovi AB, Somaschini A, Maggioni AP; on the behalf of BRING-UP-3 Heart Failure Investigators. Medical Treatments in Patients With Ambulatory Heart Failure: First Data From the BRING-UP-3 Heart Failure Study. J Card Fail. 2025 Dec;31(12):1847-1857. doi: 10.1016/j.cardfail.2025.02.019. Epub 2025 Mar 20. PMID 40118200